CLINICAL TRIAL: NCT06170047
Title: The Chicago Parent Program for Foster Care: A Randomized Control Trial Examining the Prevention of Behavior Problems Among Young Children in Foster Care Through Group-based Foster Caregiver Training
Brief Title: Chicago Parent Program for Foster and Kinship Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Johns Hopkins University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD105727 (NIH)
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Behavior Problem; Parenting
Keywords: Foster care; Child behavior; Parenting skills; Behavioral health; Prevention; Parenting confidence; Parenting stress
MeSH Terms: conditions — Mental Disorders; Child Behavior

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Principal Investigator, Co-Investigators, Statistician, and the Clinical Research Coordinator conducting the caregiver-youth DPICS observation recording and coding will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chicago Parent Program for Foster Care (Experimental): The Chicago Parent Program for Foster Care (CPP-FC) is a caregiver-directed prevention program to strengthen parenting skills and confidence in foster and kinship caregivers and prevent or reduce behavior problems in children 2-8 years old. CPP-FC was designed to specifically meet the unique needs of children ages 2-8 who are placed with foster and kinship caregivers. Participants assigned to CPP-FC will receive CPP-FC and the services typically offered from the county, Cincinnati Children's Hospital Medical Center Comprehensive Health Evaluations for Cincinnati's Kids (CHECK) clinic, and for licensed caregivers, their licensing agency.
  Interventions: Behavioral: Chicago Parent Program for Foster Care
- Usual Care (Active Comparator): Usual Care control will receive standard care offered from the county, Cincinnati Children's Hospital Medical Center Comprehensive Health Evaluations for Cincinnati's Kids (CHECK) clinic, and for licensed caregivers, their licensing agency.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Chicago Parent Program for Foster Care — CPP-FC consists of 12 two-hour sessions delivered virtually by two trained group leaders over 16 weeks (11 concurrent weeks, 1 one-month booster) in a group-based format. Foster and kinship caregivers of young children are systematically taught parenting skills through group discussions, videotaped vignettes, structured role play and weekly homework assignments.
  Other Names: CPP-FC; Caregivers on Point
  Arms: Chicago Parent Program for Foster Care
Other: Usual Care — The Usual Care control will receive services from the county, CHECK clinic, and for licensed caregivers, their licensing agency per usual care. Caregivers receive training and support from their county and/or private licensing agency, children are referred to community services by the caseworker when behaviors emerge, and support from behavioral health specialists is available when caregivers request them.
  Arms: Usual Care

SUMMARY:
The primary objective of this study is to test the effects of an evidence-based prevention intervention (CPP) adapted for foster and kinship caregivers of young children (FC; foster care) on caregiver competence and child behavior problems for children in foster care compared with an active comparator group that receives standard supports through the child welfare and healthcare systems (i.e., usual care).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the impact of an evidence-based parenting program, The Chicago Parent Program (CPP) adapted for foster and kinship caregivers of young children (CPP-FC). A parallel, two-arm, randomized controlled trial of 300 caregiver-youth dyads will be conducted, comparing the impact of CPP-FC versus a usual care control on caregivers and foster youth. Quantitative and qualitative data about CPP-FC will be collected from foster and kinship caregivers and through observations of caregivers and youth. The findings from this study will demonstrate whether CPP-FC is effective in reducing behavior problems in young foster children and whether that contributes to reduced caregiver stress, increased caregiver confidence, increased positive parenting behavior, and longer lengths of time that children remain with foster and kinship caregivers, preventing unnecessary moves from one caregiver to another and improving child wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Must be a licensed foster caregiver or kinship caregiver to a foster child between the ages of 2 and less than 9 years of age
* Must be a licensed foster caregiver or kinship caregiver to a foster child in Ohio and in the custody of Hamilton County Job and Family Services, Butler County Children Services, or Montgomery County Children Services
* Must be in good standing with the foster care agency
* Must be English-speaking

Exclusion Criteria:

* Not having a foster child between the ages of 2 and less than 9 years
* The foster child not being in the custody of Ohio counties: Hamilton County Job and Family Services, Butler County Children Services, or Montgomery County Children Services
* The foster child was placed in the home more than 45 days prior to enrollment
* The foster child being moved out of the placement prior to the start of the intervention
* The foster child having been previously enrolled with another caregiver
* The caregiver having been previously enrolled with another child
* The caregiver unable to commit to completing all study activities
* The foster child is not enrolled in the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Stress Scale | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Parental Stress Scale is an 18-item questionnaire that assesses parental stress relating to parental sensitivity to the child, child behavior, and quality of the caregiver-child relationship. Items are rated on a 5-point scale, ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Some items are reverse scored. Items are summed to yield a total score, with higher scores indicating higher levels of parental stress.
Change in Perceived Stress Scale | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Perceived Stress Scale is a 14-item self-report measure of how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. All items are rated on a 5-point scale, ranging from 0 ("Never") to 4 ("very often"). Some items are reverse scored. Responses are summed to yield a total score (range 0-56), with higher scores indicating greater perceived stress.
The Child Adjustment & Parent Efficacy Scale, Total Intensity subscale | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Child Adjustment & Parent Efficacy Scale, Total Intensity subscale is a 27-item measure of child behavior and emotional problems. Item responses are rated on a 4-point scale, ranging from 0 ("Not true of my child at all") to 3 ("True of my child very much"/"Most of the time"). Twenty-four items are summed to yield a Behavior Problems score (range 0-72), and three items are summed to yield an Emotional Problems score (range 0-9). Behavioral and Emotional Problems scores can be summed for a Total Intensity score (range 0-81). Higher scores indicate a higher level of problems.
The Child Adjustment & Parent Efficacy Scale, Parenting Efficacy subscale | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Child Adjustment & Parent Efficacy Scale, Parenting Efficacy subscale is a 19-item measure of parental self-efficacy. Item responses are rated on a 10-point scale, with responses ranging from 1 ("Certain I can't do it") to 10 ("Certain I can do it"). Items are summed to yield a total efficacy score, with higher scores indicating higher self-efficacy.
Change in Parenting Sense of Competence Scale | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Parenting Sense of Competence Scale is a 17-item questionnaire that measures overall parenting satisfaction and competence. Items are measured on a 6-point scale, with responses ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). Some items are reverse scored. Items are summed to yield two subscales: parental satisfaction and parental self-efficacy. Higher scores indicate higher levels of parental satisfaction and parental self-efficacy.

SECONDARY OUTCOMES:
Change in Parenting Behaviors and Dimensions Questionnaire | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Parenting Behaviors and Dimensions Questionnaire is a 33-item measure of contemporary parenting behavior that measures six core dimensions of parenting: Emotional Warmth, Punitive Discipline, Anxious Intrusiveness, Autonomy Support, Permissive Discipline, and Democratic Discipline. Items are rated on a 6-point scale ranging from 1 ("Never") to 7 ("Always"). Higher scores indicate higher levels of the parenting dimension.
Change in child behavior | Baseline, 3 months (mid-point), and 6 months (follow-up)
  The Strengths and Difficulties Questionnaire is a 25-item questionnaire that assesses child behavior. Items are rated on a 3-point scale and responses range from 0 ("Not true") to 2 ("Certainly true"). Some items are reverse scored. Items are summed to yield 5 subscales: Emotional Problems, Conduct Problems, Hyperactivity, Peer Problems, and Prosocial. A total score is calculated using the sum of all the subscales, except Prosocial. Higher scores in each subscale and the total score indicate more child behavior problems.
Change in child self-regulation | Baseline and 3 months
  A 5-minute caregiver-child behavioral observation will be recorded and subsequently coded by two trained coordinators and the PI using is the Dyadic Parent-Child Interaction Coding System Comprehensive Manual for Research and Training 4th edition (DPICS-IV).91 The observation will involve a free-play period and a caregiver-directed clean-up from the play activity. The recording will be coded for caregiver positive statements (acknowledgment, description, unlabeled praise, labeled praise, reflection), statements to avoid (questions, indirect commands, negative talk), and direct commands. Child compliance, non-compliance, and instances where the child did not have the opportunity to comply with caregiver commands are also coded.
Number of children experiencing placement change due to child behavior problems. | 12 months
  The child welfare administrative record will be reviewed to assess number of child participants experiencing a placement change due to child behavior problems.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Beal, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the open science movement and with the directive of clinicaltrials.gov to include a data sharing plan in submissions, we will have the following data sharing policy: we will share with other investigators (1) all individual participant data after deidentification, and (2) study management documents (protocol, statistical analysis plan, consent form, analytic code, data dictionary).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: These will be made available three months after publication of the primary article and ending five years after publication.
Access Criteria: Those requesting data will be required to submit a proposal to the PI. This will be reviewed by the investigative team for methodological soundness and scientific merit. Proposals approved by the PI will be shared with the legal department at Cincinnati Children's Hospital Medical Center and prosecuting attorneys and directors of children's services at Hamilton, Butler, and Montgomery counties for approval. Once approved by all parties, a data use agreement will be established with the outside investigator before data is shared. This plan is consistent with guidelines developed by the International Committee of Medical Journal Editors (Taichman,D S, et. al, 2017) and established memoranda of understanding between Cincinnati Children's and children's services agencies for research involving children in foster and kinship care.

REFERENCES:
- [Background] Berry, J. O., & Jones, W. H. (1995). The parental stress scale: Initial psychometric evidence. Journal of Social and Personal Relationships, 12, 463-472. http://dx.doi.org/10.1177/0265407595123009
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gibaud-Wallston J, Wandersman LP. Parenting Sense of Competence Scale. Lawrence Erlbaum Associates.; 1978. Accessed October 13, 2021. https://www.bristol.ac.uk/media-
- [Background] Reid CA, Roberts LD, Roberts CM, Piek JP. Towards a model of contemporary parenting: the parenting behaviours and dimensions questionnaire. PLoS One. 2015 Jun 4;10(6):e0114179. doi: 10.1371/journal.pone.0114179. eCollection 2015. PMID 26043107
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Research and Training DPICS-IV Manual (2013). PCIT. Accessed October 5, 2021. http://www.pcit.org/store/p19/Research_and_Training_DPICS-IV_Manual_%282013%29.html
- [Background] Taichman DB, Sahni P, Pinborg A, Peiperl L, Laine C, James A, Hong ST, Haileamlak A, Gollogly L, Godlee F, Frizelle FA, Florenzano F, Drazen JM, Bauchner H, Baethge C, Backus J. Data Sharing Statements for Clinical Trials: A Requirement of the International Committee of Medical Journal Editors. Ann Intern Med. 2017 Jul 4;167(1):63-65. doi: 10.7326/M17-1028. Epub 2017 Jun 6. No abstract available. PMID 28586790
- [Background] Alina Morawska, Matthew R Sanders, Divna Haslam, Ania Filus & Renee Fletcher (2014) Child Adjustment and Parent Efficacy Scale: Development and Initial Validation of a Parent Report Measure, Australian Psychologist, 49:4, 241-252, DOI: 10.1111/ap.12057
- [Derived] Beal SJ, Zion C, Mara CA, Patel MA, Bettencourt AF, Breitenstein SM, Vaughn LM, Greiner MV, Ammerman RT. Caregivers on point: a randomized treatment-control prevention trial for foster and kinship caregivers to reduce behavior challenges among children in foster care. Trials. 2024 Oct 10;25(1):670. doi: 10.1186/s13063-024-08524-9. PMID 39390601